CLINICAL TRIAL: NCT03276936
Title: An Open-Label Study to Evaluate the Long-Term Safety of Topical Administration of FMX103 for 40 Weeks in the Treatment of Moderate to Severe Facial Papulopustular Rosacea (Study FX2016-13)
Brief Title: A Study to Evaluate the Long-Term Safety of Topical Administration of FMX103 in the Treatment of Moderate to Severe Papulopustular Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX2016-13
Record Dates: First submitted 2017-08-21; First posted 2017-09-08 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Minocycline Foam 1.5% (Experimental): FMX-103
  Interventions: Drug: FMX103 1.5%

INTERVENTIONS:
Drug: FMX103 1.5% — FMX103 1.5% minocycline foam

SUMMARY:
The primary objective is to show that open-label extended treatment with FMX103 1.5%, for up to an additional 40 weeks, is safe and well tolerated.

DETAILED DESCRIPTION:
This is an open-label, multicenter, 40-week extension study to evaluate the long-term safety, tolerability, and efficacy of FMX103 1.5% topical foam in the treatment of moderate-to-severe facial papulopustular rosacea. Subjects entering this study will have recently participated in 1 of 2 pivotal, double-blind, vehicle-controlled, safety and efficacy studies (FX2016-11 and FX2016-12 - NCT03142451). Subjects must demonstrate that they are eligible to continue into Study FX2016-13 based on safety evaluations and IGA score performed at Final Visit of one of the previous double-blind studies.

At the completion of the Final Visit in Study FX2016-11 or Study FX2016-12, subjects may be invited to continue into this open-label study for an additional 40 weeks of open-label treatment. A minimum of 400 subjects will be enrolled into from Studies FX2016-11 and FX2016-12. Subjects who elect to continue into this open-label study will receive supplies of active FMX103 1.5% minocycline foam.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed 12 weeks of treatment in either Study FX2016-11 or Study FX2016-12.
2. Have not had a worsening of disease, determined by the Investigator's Global Assessment (IGA), at Visit 5/Week 12 (Final Visit) relative to the Day 0/Baseline assessment in Study FX2016-11 or Study FX2016-12.

Exclusion Criteria:

1. Have a new systemic disease or condition, including an ongoing AE that might interfere with the conduct of the study or the interpretation of results.
2. Have developed a condition that would have been exclusionary for Study FX2016-11 or Study FX2016-12, including pseudomembranous colitis, antibiotic associated colitis, hepatitis, liver damage, renal impairment, drug addiction, or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (79):
  - Foamix Investigational Site # 207, Glendale, Arizona
  - Foamix Investigational Site # 202, Hot Springs, Arkansas
  - Foamix Investigational Site # 222, Rogers, Arkansas
  - Foamix Investigational Site # 127, Fremont, California
  - Foamix Investigational Site # 226, Los Angeles, California
  - Foamix Investigational Site # 220, Murrieta, California
  - Foamix Investigational Site # 131, Oceanside, California
  - Foamix Investigational Site # 134, Sacramento, California
  - Foamix Investigational Site # 114, San Diego, California
  - Foamix Investigational Site # 116, San Luis Obispo, California
  - Foamix Investigational Site # 135, Santa Ana, California
  - Foamix Investigational Site # 123, Santa Monica, California
  - Foamix Investigational Site # 239, Temecula, California
  - Foamix Investigational Site # 227, Denver, Colorado
  - Foamix Investigational Site # 223, Boca Raton, Florida
  - Foamix Investigational Site # 215, Boynton Beach, Florida
  - Foamix Investigational Site # 109, Clearwater, Florida
  - Foamix Investigational Site # 240, Fort Myers, Florida
  - Foamix Investigational Site # 112, Hialeah, Florida
  - Foamix Investigational Site # 214, Miami, Florida
  - Foamix Investigational Site # 241, North Miami Beach, Florida
  - Foamix Investigational Site # 104, Ormond Beach, Florida
  - Foamix Investigational Site # 121, Sanford, Florida
  - Foamix Investigational Site # 125, Tampa, Florida
  - Foamix Investigational Site # 124, West Palm Beach, Florida
  - Foamix Investigational Site # 118, Alpharetta, Georgia
  - Foamix Investigational Site # 204, Newnan, Georgia
  - Foamix Investigational Site # 233, Sandy Springs, Georgia
  - Foamix Investigational Site # 139, Snellville, Georgia
  - Foamix Investigational Site # 211, Arlington Heights, Illinois
  - Foamix Investigational Site # 138, New Albany, Indiana
  - Foamix Investigational Site # 225, Newburgh, Indiana
  - Foamix Investigational Site # 218, South Bend, Indiana
  - Foamix Investigational Site # 235, Louisville, Kentucky
  - Foamix Investigational Site # 237, Louisville, Kentucky
  - Foamix Investigational Site # 102, Metairie, Louisiana
  - Foamix Investigational Site # 115, New Orleans, Louisiana
  - Foamix Investigational Site # 110, Beverly, Massachusetts
  - Foamix Investigational Site # 107, Brighton, Massachusetts
  - Foamix Investigational Site # 229, Watertown, Massachusetts
  - Foamix Investigational Site # 137, Ann Arbor, Michigan
  - Foamix Investigational Site # 242, Bay City, Michigan
  - Foamix Investigational Site # 210, Detroit, Michigan
  - Foamix Investigational Site # 103, Fort Gratiot, Michigan
  - Foamix Investigational Site # 120, Troy, Michigan
  - Foamix Investigational Site # 140, Warren, Michigan
  - Foamix Investigational Site # 232, Fridley, Minnesota
  - Foamix Investigational Site # 130, Saint Joseph, Missouri
  - Foamix Investigational Site # 133, Omaha, Nebraska
  - Foamix Investigational Site # 221, Las Vegas, Nevada
  - Foamix Investigational Site # 136, New York, New York
  - Foamix Investigational Site # 111, Stony Brook, New York
  - Foamix Investigational Site # 119, Charlotte, North Carolina
  - Foamix Investigational Site # 238, High Point, North Carolina
  - Foamix Investigational Site # 212, Raleigh, North Carolina
  - Foamix Investigational Site # 234, Winston-Salem, North Carolina
  - Foamix Investigational Site # 101, Bexley, Ohio
  - Foamix Investigational Site # 128, Dublin, Ohio
  - Foamix Investigational Site # 236, Norman, Oklahoma
  - Foamix Investigational Site # 224, Exton, Pennsylvania
  - Foamix Investigational Site # 141, Jenkintown, Pennsylvania
  - Foamix Investigational Site # 129, Yardley, Pennsylvania
  - Foamix Investigational Site # 105, Johnston, Rhode Island
  - Foamix Investigational Site # 231, Charleston, South Carolina
  - Foamix Investigational Site # 106, Greenville, South Carolina
  - Foamix Investigational Site # 230, Mt. Pleasant, South Carolina
  - Foamix Investigational Site # 228, Knoxville, Tennessee
  - Foamix Investigational Site # 219, Arlington, Texas
  - Foamix Investigational Site # 132, Austin, Texas
  - Foamix Investigational Site # 117, Austin, Texas
  - Foamix Investigational Site # 201, Houston, Texas
  - Foamix Investigational Site # 206, Pflugerville, Texas
  - Foamix Investigational Site # 108, San Antonio, Texas
  - Foamix Investigational Site # 208, San Antonio, Texas
  - Foamix Investigational Site # 213, San Antonio, Texas
  - Foamix Investigational Site # 209, Webster, Texas
  - Foamix Investigational Site # 126, Salt Lake City, Utah
  - Foamix Investigational Site # 216, Lynchburg, Virginia
  - Foamix Investigational Site # 203, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://foamix.co.il/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, multi-center, 40-week extension study was conducted at 70 sites in the United States from 05 September 2017 to 03 January 2019, and enrolled participants from previous double-blind (DB) studies FX2016-11 and FX2016-12.
Pre-assignment Details: Baseline for the study was conducted at the same time as Visit 5/Week 12 (Final Visit) of Study FX2016-11 or Study FX2016-12. All assessments performed at Visit 5/Week 12 (Final Visit) of Study FX2016-11 or Study FX2016-12 were not repeated but rather recorded as the same assessments at Baseline for this study.
Groups:
- DB-FMX103 1.5% Minocycline Foam; DB-Vehicle Foam: Enrolled participants from Study FX2016-11 and Study FX2016-12 (FMX103 1.5% group) applied FMX103 1.5% minocycline foam topically to the face once daily for 40 weeks in this present Study FX2016-13. Participants were grouped based on their experience in the previous double-blind study, and that all participants received the study drug in an open-label fashion.
Period: Overall Study
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Started | 332 | 172
Completed | 276 | 134
Not Completed | 56 | 38
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 16 | 13
Not completed — Withdrawal by Subject | 30 | 20
Not completed — Not mentioned | 6 | 3

BASELINE CHARACTERISTICS:
Population: All treated population included all participants who used the study drug at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam | Total
Number analyzed (Participants) | 332 | 172 | 504
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (12.62) | 51.9 (11.90) | 51.4 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 110 | 351
  Male | 91 | 62 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 31 | 93
  Not Hispanic or Latino | 269 | 141 | 410
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 321 | 163 | 484
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Inflammatory Lesion Count at Week 40
Description: Change from Baseline (Baseline visit in the initial DB study [FX2016-11 or FX2016-12] and Baseline visit of the open-label extension study [Week 12]) in inflammatory lesion count at Week 40 is reported. The lesion counts performed at Week 12 [Final Visit] in Study FX2016-11 or Study FX2016-12 constituted as the Baseline value for this study. Changes from Baseline were calculated as the Baseline [pre-dose] value minus the post-Baseline value, so that decreases reflected a reduction in lesion count. The number of papules, pustules, and nodules were counted, and the numbers recorded.
Time Frame: Day 0/ Baseline (Final visit of previous DB study [Week 12]) and at Week 40
Population: All treated population included all participants who used the study drug at least once. Here, overall number of participants analyzed (N) signifies only the participants with available data that were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 272 | 129
Lesions | 23.0 (10.96) | 22.5 (10.83)

2. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessments (IGA) Treatment Success at Week 40
Description: The IGA scale for Rosacea, was used by the Investigators to assess the severity of a participant's Rosacea. The scale ranges from 0 (Clear): No inflammatory papules or pustules to 4 (Severe): Many inflammatory papules or pustules, and up to 2 nodules. Higher scores indicated severe outcome. Treatment success was defined as an IGA score of 0 (score of clear) or 1 (almost clear), and at least a 2-grade improvement (decrease) from Baseline.
Time Frame: At Week 40
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 272 | 129
Percentage of participants | 81.6 | 76.0

3. Secondary Outcome: Absolute Change From Baseline in Inflammatory Lesion Count at Weeks 4, 10, 16, 22, 28, and 34
Description: as for outcome 1
Time Frame: Day 0/ Baseline (Final visit of previous DB study [Week 12]) and at Weeks 4, 10, 16, 22, 28, and 34
Population: All treated population included all participants who used the study drug at least once. Here, number analyzed (n) signifies only the participants with available data that were analyzed at given specified week.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 332 | 172
Lesions
  Week 4: number analyzed (Participants) | 326 | 168
  Week 4 | 19.5 (11.57) | 17.4 (12.18)
  Week 10: number analyzed (Participants) | 321 | 156
  Week 10 | 20.4 (11.62) | 19.8 (12.92)
  Week 16: number analyzed (Participants) | 310 | 150
  Week 16 | 21.9 (11.38) | 20.0 (13.09)
  Week 22: number analyzed (Participants) | 298 | 146
  Week 22 | 22.2 (12.35) | 20.7 (11.33)
  Week 28: number analyzed (Participants) | 286 | 138
  Week 28 | 22.4 (11.89) | 21.7 (10.89)
  Week 34: number analyzed (Participants) | 279 | 136
  Week 34 | 23.2 (11.75) | 22.5 (10.71)

4. Secondary Outcome: Percentage of Participants Achieving IGA Treatment Success at Weeks 4, 10, 16, 22, 28 and 34
Description: as for outcome 2
Time Frame: At Weeks 4, 10, 16, 22, 28 and Week 34
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 332 | 172
Percentage of participants
  Week 4: number analyzed (Participants) | 326 | 168
  Week 4 | 50.6 | 48.2
  Week 10: number analyzed (Participants) | 321 | 156
  Week 10 | 60.1 | 54.5
  Week 16: number analyzed (Participants) | 310 | 150
  Week 16 | 68.1 | 64.0
  Week 22: number analyzed (Participants) | 298 | 146
  Week 22 | 69.1 | 64.4
  Week 28: number analyzed (Participants) | 286 | 138
  Week 28 | 72.4 | 65.9
  Week 34: number analyzed (Participants) | 279 | 136
  Week 34 | 73.5 | 72.1

5. Secondary Outcome: Percentage Change From Baseline in Inflammatory Lesion Count at Weeks 4, 10, 16, 22, 28, and 34
Description: as for outcome 1
Time Frame: Day 0/ Baseline (Final visit of previous DB study [Week 12]) and at Weeks 4, 10, 16, 22, 28, and 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 332 | 172
Percent Change
  Week 4: number analyzed (Participants) | 326 | 168
  Week 4 | 67.91 (27.569) | 61.25 (32.306)
  Week 10: number analyzed (Participants) | 321 | 156
  Week 10 | 72.43 (27.937) | 69.02 (32.966)
  Week 16: number analyzed (Participants) | 310 | 150
  Week 16 | 77.36 (22.739) | 71.46 (33.230)
  Week 22: number analyzed (Participants) | 298 | 146
  Week 22 | 77.51 (25.101) | 73.63 (27.515)
  Week 28: number analyzed (Participants) | 286 | 138
  Week 28 | 78.82 (23.439) | 77.06 (25.863)
  Week 34: number analyzed (Participants) | 279 | 136
  Week 34 | 81.91 (20.549) | 80.38 (22.873)

6. Secondary Outcome: Number of Participants Reporting Satisfaction and Dissatisfaction With the Study Drug Based on Subject Satisfaction Questionnaire (SSQ) at Week 40
Description: The questionnaire consisted of questions with responses on scale with scores: as 1 (Very satisfied or Very likely ) to 5 (Very dissatisfied or Very unlikely) for each variable as for example, Easy to use, 1 is very satisfied and 5 is very dissatisfied. The minimum score represented best outcome and higher score represented worst outcome.
Time Frame: At Week 40
Population: All treated population included all participants who used the study drug at least once. Here, number analyzed are number of participants analyzed for given variable.
Measure: Number; unit: Participants
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 332 | 172
Participants
  Easy to Use; 1-Very satisfied: number analyzed (Participants) | 266 | 128
  Easy to Use; 1-Very satisfied | 178 | 82
  Easy to Use; 5-Very dissatisfied: number analyzed (Participants) | 266 | 128
  Easy to Use; 5-Very dissatisfied | 0 | 2
  Feel on Skin; 1-Very satisfied: number analyzed (Participants) | 266 | 128
  Feel on Skin; 1-Very satisfied | 110 | 47
  Feel on Skin; 5-Very dissatisfied: number analyzed (Participants) | 266 | 128
  Feel on Skin; 5-Very dissatisfied | 3 | 3
  Odor; 1-Very satisfied: number analyzed (Participants) | 266 | 128
  Odor; 1-Very satisfied | 155 | 78
  Odor; 5-Very dissatisfied: number analyzed (Participants) | 266 | 128
  Odor; 5-Very dissatisfied | 0 | 0
  Color; 1-Very satisfied: number analyzed (Participants) | 266 | 128
  Color; 1-Very satisfied | 107 | 44
  Color; 5-Very dissatisfied: number analyzed (Participants) | 266 | 128
  Color; 5-Very dissatisfied | 10 | 7
  Ease of application; 1-Very satisfied: number analyzed (Participants) | 266 | 128
  Ease of application; 1-Very satisfied | 183 | 88
  Ease of application; 5-Very dissatisfied: number analyzed (Participants) | 266 | 128
  Ease of application; 5-Very dissatisfied | 0 | 0
  Ease fitting in to daily routine; 1-Very satisfied: number analyzed (Participants) | 266 | 128
  Ease fitting in to daily routine; 1-Very satisfied | 155 | 83
  Ease fitting in to daily routine; 5-Very dissatisfied: number analyzed (Participants) | 266 | 128
  Ease fitting in to daily routine; 5-Very dissatisfied | 0 | 0
  Compared to Other Products;1-Very satisfied: number analyzed (Participants) | 265 | 127
  Compared to Other Products;1-Very satisfied | 144 | 70
  Compared to Other Products; 5-Very dissatisfied: number analyzed (Participants) | 265 | 127
  Compared to Other Products; 5-Very dissatisfied | 1 | 2
  Use with other rosacea treatments; 1-Very likely: number analyzed (Participants) | 266 | 127
  Use with other rosacea treatments; 1-Very likely | 153 | 74
  Use with other rosacea treatments; 5-Very unlikely: number analyzed (Participants) | 266 | 127
  Use with other rosacea treatments; 5-Very unlikely | 3 | 5
  Recommend to friend; 1-Very likely: number analyzed (Participants) | 265 | 128
  Recommend to friend; 1-Very likely | 156 | 75
  Recommend to friend; 5-Very unlikely: number analyzed (Participants) | 265 | 128
  Recommend to friend; 5-Very unlikely | 3 | 1
  Overall Satisfaction with Product; 1-Very satisfied: number analyzed (Participants) | 265 | 128
  Overall Satisfaction with Product; 1-Very satisfied | 155 | 75
  Overall Satisfaction with Product; 5-Very dissatisfied: number analyzed (Participants) | 265 | 172
  Overall Satisfaction with Product; 5-Very dissatisfied | 2 | 1

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Evaluation of the long-term safety of topical FMX103 1.5% minocycline foam in the treatment of moderate to severe facial papulopustular rosacea for 40 weeks. A Treatment-emergent Adverse Events (TEAEs) was defined as any AE with an onset date after the first dose date of the open-label extension study and before the last application of study drug plus 3 days having been absent pre-treatment or worsened relative to the pre-treatment state.
Time Frame: Day 0/ Baseline (Final visit of previous DB study [Week 12]) until safety follow-up (Week 44)
Population: All treated population included all participants who used the study drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | DB-FMX103 1.5% Minocycline Foam | DB-Vehicle Foam
Number analyzed (Participants) | 332 | 172
Participants
  All AEs | 151 | 70
  TEAEs | 137 | 64
  Serious TEAEs | 9 | 4
  Treatment-related TEAEs | 5 | 8
  Adverse events leading to study discontinuation | 3 | 2
  Participants with any severe TEAE | 6 | 6
  Death | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 0/ Baseline (Final visit of previous DB study [Week 12]) until safety follow-up (Week 44)
Groups:
- Minocycline Foam 1.5%: Participants applied FMX103 1.5% minocycline foam topically to the face once daily for 40 weeks.
- Vehicle Foam: Participants applied matching vehicle foam topically to the face once daily for 40 weeks.
Arm/Group | Minocycline Foam 1.5% | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 1/332 | 0/172
Serious Adverse Events (participants affected / at risk) | 9/332 | 4/172
Other Adverse Events (participants affected / at risk) | 8/332 | 11/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline Foam 1.5% (N=332) | Vehicle Foam (N=172)
Appendicitis perforated (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline Foam 1.5% (N=332) | Vehicle Foam (N=172)
Sinusitis (Infections and infestations) | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT03276936/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT03276936/SAP_001.pdf